CLINICAL TRIAL: NCT06329947
Title: A Phase II Study of Surufatinib Combined With Camrelizumab and mFOLFOX6 as Second-line Treatment for Advanced PRAD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rui-hua Xu, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Rui-hua Xu, MD, PhD, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-P106
Record Dates: First submitted 2023-12-05; First posted 2024-03-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — surufatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Surufatinib in combination with Camrelizumab and mFOLFOX6
  Interventions: Drug: Surufatinib 250mg/d qd once daily

INTERVENTIONS:
Drug: Surufatinib 250mg/d qd once daily — mFOLFOX6( Oxaliplatin + Leucovorin + fluorouracil) Oxaliplatin 85mg/m2 d1+CF 400mg/m2 d1+5-FU 400mg/m2d1 /2400mg/m2 continuous intravenous injection (civ) for 46h, The drug is administered every 14 days for a total of 8-12 cycles.
  Other Names: Camrelizumab 200mg,IV,Q2W once every 21 days during the maintenance treatment period, for a maximum of 2 years

SUMMARY:
To preliminarily evaluate whether there is a survival benefit of surufatinib combined with camrelizumab and mFOLFOX6 as the second-line treatment for advanced pancreatic cancer, and to explore the feasibility of second-line and post-line treatment for advanced pancreatic cancer

DETAILED DESCRIPTION:
Second-line clinical study of surufatinib in combination with Caralizumab advanced pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. Have full understanding of this study and voluntarily sign the informed consent form;
2. Male and Female aged between 18 and 75 years are eligible;
3. Histologically or cytologically confirmed metastatic pancreatic cancer;
4. Patients who have previously failed first-line gemcitabine-based chemotherapy or have disease progression/recurrence during previous neoadjuvant/adjuvant treatment or within 6 months after the end of treatment are considered to have failed first-line systemic chemotherapy; neoadjuvant/adjuvant treatment plan Also gemcitabine-based chemotherapy;
5. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
7. Predicted survival ≥12 weeks;
8. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Participated in other anti-tumor drug clinical trials within 28 days;
2. Have previously received any anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody or acted on T cell costimulation or checkpoints Treatment with any other antibodies of the pathway (such as OX40, CD137, etc.);
3. Have previously received anti-vascular endothelial growth factor/vascular endothelial growth factor receptor (VEGF/VEGFR) targeted drug treatment;
4. Those who are known to be allergic to any of the drugs in the study;
5. Brain metastasis accompanied by symptoms or symptom control time <2 months;
6. The subject has suffered from other malignant tumors in the past or at the same time within 5 years (except cured basal cell carcinoma of the skin and cervical cancer in situ);
7. Insufficient bone marrow hematopoietic function (without blood transfusion within 14 days):

   1. Absolute neutrophil count (ANC) <1.5×109/L;
   2. Platelets <100×109/L;
   3. Hemoglobin <8g/dL.
8. Liver abnormalities:

   1. When there is no liver metastasis, ALT, AST or ALP>2.5×the upper limit of the normal reference range (ULN); when there is liver metastasis, ALT, AST or ALP>5×ULN;
   2. Serum total bilirubin >1.5×ULN (Gilber syndrome >3×ULN);
   3. Decompensated cirrhosis (Child-Pugh liver function grade B or C);
   4. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA copy number ≥2000IU/mL (those who are HBsAg positive and hepatitis B virus DNA copy number <2000IU/mL need to receive at least 2 weeks of anti-HBV treatment before taking the first dose) ;
   5. Hepatitis C virus (HCV) antibody positive and HCVRNA test positive.
9. Kidney abnormalities:

   1. Serum creatinine>1.5×ULN;
   2. Routine urine test shows urine protein ≥++, and the 24-hour urine protein quantification is confirmed to be >1.0g;
   3. Renal failure requiring hemodialysis or peritoneal dialysis;
   4. Past history of nephrotic syndrome.；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-05-22 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Time Frame: up to 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
disease control rate (DCR) | Time Frame: up to 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | Time Frame: up to 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
overall survival (OS) | Time Frame: up to 24 months
  OS is the time from enrollment to death due to any cause.
quality of life (QoL) | Time Frame: up to 24 months
  Assessing the quality of life of cancer patients by QLQ-C30
adverse events (AE) | Time Frame: up to 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Hua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- SunYat-senUniversity Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT06329947/Prot_000.pdf
  • Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT06329947/ICF_001.pdf